CLINICAL TRIAL: NCT07248475
Title: Effects of Battle Rope Training on ROM and Pain in Children With Post Traumatic Elbow Contractures.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/Azlfakarim
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Children, Adult
Keywords: Battle Rope Training; Elbow Contractures; ROM
MeSH Terms: interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: n this randomized controlled trial, participants will be divided into two groups: a control group, receiving standard treatment (ROM exercises, stretching, and heat therapy), and an intervention group, receiving the same standard treatment plus battle rope training. ROM exercises and stretching will focus on gentle elbow flexion and extension to enhance flexibility, while heat therapy will prepare muscles for movement.
  The intervention group will additionally perform 10-15 minutes of battle rope training, involving dynamic movements that engage the upper body and increase joint activation
Who Masked: Participant
Masking Description: Participant will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Battle Rope Training (Active Comparator): Group A will perform Baseline treatment with Battle rope trining.The intervention group will follow the same baseline rehabilitation program of ROM exercises, stretching, and heat therapy as the control group to ensure a consistent foundation for all participants. However, in addition to these therapies, the intervention group will engage in Battle Rope Training designed to further enhance muscle activation, endurance, and joint mobility. All five exercises will be performed 5 days a week with 2 sets.A 12.8-m TR (4.1 kg) was used for all trials.
  Interventions: Other: Battle Rope Training
- ROM, Stretching and Heat Therapy (Active Comparator): The control group will receive Range of Motion (ROM) exercises, stretching, and heat therapy to manage post-traumatic elbow contracture. ROM Exercises will focus on gentle flexion and extension movements to gradually improve joint mobility . These exercises will be performed daily.Stretching exercises will target the muscles surrounding the elbow specifically designed to lengthen and relax the soft tissues that may contribute to contracture. These stretches will be held for 15-30 seconds and repeated several times per session to facilitate flexibility without overstressing the joint. Heat Therapy will be applied to the affected area . Heat will be applied for approximately 10-15 minutes. This combined approach aims to provide standard care that helps alleviate stiffness, manage pain, and improve functional movement over time, without the addition of the battle rope intervention
  Interventions: Other: Stretching and Heat Therapy

INTERVENTIONS:
Other: Battle Rope Training — All five exercises will be performed 5 days a week with 2 sets.A 12.8-m TR (4.1 kg) was used for all trials Week 1 to 2: During the period the subjects performed 5 selected battle rope exercises. Each exercises the subjects performed ten seconds with two repetitions. The total number of set was 2. The recovery for in between exercise 1minute and in between set was 5 minutes. Week 3 to 4: During the period the subjects performed 5 selected battle rope exercises. Each exercises the subjects performed twenty seconds with 3 repetitions. The total number of set was 2. The recovery for in between exercise 1minute and in between set was 5 minutes. Week 5 to 6: During the period the subjects performed 5 selected battle rope exercises. Each exercises the subjects performed thirty seconds with 4 repetitions. The total number of set was 2. The recovery for in between exercise 1minute and in between set was 5 minutes
  Arms: Battle Rope Training
Other: Stretching and Heat Therapy — The control group will receive Range of Motion (ROM) exercises, stretching, and heat therapy to manage post-traumatic elbow contracture. ROM Exercises will focus on gentle flexion and extension movements to gradually improve joint mobility . These exercises will be performed daily.Stretching exercises will target the muscles surrounding the elbow specifically designed to lengthen and relax the soft tissues that may contribute to contracture. These stretches will be held for 15-30 seconds and repeated several times per session to facilitate flexibility without overstressing the joint. Heat Therapy will be applied to the affected area . Heat will be applied for approximately 10-15 minutes. This combined approach aims to provide standard care that helps alleviate stiffness, manage pain, and improve functional movement over time, without the addition of the battle rope intervention
  Arms: ROM, Stretching and Heat Therapy

SUMMARY:
The primary objective of this study is to assess the effectiveness of battle rope training in improving ROM, reducing pain, and enhancing overall elbow function in children with post-traumatic elbow contracture. By comparing standard therapy alone to standard therapy plus battle rope training, the study aims to determine if this added intervention leads to greater improvements in functional mobility and pain relief.In this randomized controlled trial, participants will be divided into two groups: a control group, receiving standard treatment (ROM exercises, stretching, and heat therapy), and an intervention group, receiving the same standard treatment plus battle rope training. ROM exercises and stretching will focus on gentle elbow flexion and extension to enhance flexibility, while heat therapy will prepare muscles for movement.

The intervention group will additionally perform 10-15 minutes of battle rope training, involving dynamic movements that engage the upper body and increase joint activation. Pre- and post-intervention assessments using a goniometer for ROM, the Flynn scoring system for functional and cosmetic outcomes, and the Visual Analogue Scale (VAS) for pain will provide comprehensive data on the effectiveness of the intervention

DETAILED DESCRIPTION:
Post-traumatic elbow contracture is a common condition in children following elbow injuries, leading to restricted range of motion (ROM), pain, and reduced arm function. Standard treatments often include stretching, heat therapy, and ROM exercises to improve joint mobility and reduce discomfort. However, new approaches such as battle rope training, which is typically used for dynamic strength and endurance, may provide additional benefits by engaging upper body muscles and enhancing functional movement in children with contractures. This study explores whether incorporating battle rope training into a standard rehabilitation program can yield better outcomes than traditional therapy alone.

The primary objective of this study is to assess the effectiveness of battle rope training in improving ROM, reducing pain, and enhancing overall elbow function in children with post-traumatic elbow contracture. By comparing standard therapy alone to standard therapy plus battle rope training, the study aims to determine if this added intervention leads to greater improvements in functional mobility and pain relief.In this randomized controlled trial, participants will be divided into two groups: a control group, receiving standard treatment (ROM exercises, stretching, and heat therapy), and an intervention group, receiving the same standard treatment plus battle rope training. ROM exercises and stretching will focus on gentle elbow flexion and extension to enhance flexibility, while heat therapy will prepare muscles for movement.

The intervention group will additionally perform 10-15 minutes of battle rope training, involving dynamic movements that engage the upper body and increase joint activation. Pre- and post-intervention assessments using a goniometer for ROM, the Flynn scoring system for functional and cosmetic outcomes, and the Visual Analogue Scale (VAS) for pain will provide comprehensive data on the effectiveness of the intervention. This study seeks to offer new insights into pediatric rehabilitation, potentially introducing an effective and engaging therapy option for managing elbow contracture in children

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to 15
* Children Suffering from Post-Traumatic Elbow Contracture
* Written informed consent obtained from the parents or guardians
* Participants must report a pain level of at least 3 on a visual analog scale (VAS)
* Children must be able to follow instructions and participate in physical activities.
* Children without any other co-existing illness like Burn Contractures
* Either gender will be included

Exclusion Criteria:

* Post Traumatic Contracture other than Elbow region
* Known allergies to materials used in battle rope training.
* Children who are unable to commit to the training schedule or follow-up assessments.
* Use of medications that may affect pain perception or muscle function, such as opioids or muscle relaxants.
* Burn Contracture.
* Presence of other significant musculoskeletal disorders or neurological conditions affecting the elbow.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1st week to 5th week
  The Visual Analogue Scale (VAS) is used to measure pain intensity in children with post-traumatic elbow contracture (17). A 10 cm line is provided, with 0 cm indicating "no pain" and 10 cm representing the "worst pain imaginable." Children are asked to mark their current pain level on this line. The distance from the "no pain" end to the mark (measured in cm) is recorded as their pain score (0-10).
  Scoring Interpretation:
  * 0 cm: No pain
  * 1-3 cm: Mild pain
  * 4-6 cm: Moderate pain
  * 7-10 cm: Severe pain VAS scores are collected before and after each intervention to track changes in pain. Lower scores over time would suggest effective pain relief from the battle rope training.
ROM using Goniometer | 1st week to 5th week
  The goniometer is a precise instrument used to measure joint angles and assess the range of motion (ROM) of the elbow(17).It will provide quantifiable data on elbow flexion and extension angles before, during, and after the intervention with battle rope training. Elbow contracture limits joint movement, so any increase in ROM captured by the goniometer can indicate a positive outcome from the intervention. For each measurement, the goniometer will be placed along the lateral aspect of the elbow, with one arm aligned along the humerus and the other along the forearm. The degree of extension and flexion will be measured in a standard position to ensure consistency across multiple sessions. The goniometer offers objective, reproducible data that will help gauge the effectiveness of battle rope training in improving joint flexibility and reducing the severity of contracture. Changes in ROM captured across the study period will be key indicators of functional improvements.
Flynn Scoring | 1st week to 5th week
  The Flynn scoring system is used to assess the functional and cosmetic outcomes in pediatric elbow injuries, providing a comprehensive score based on a range of clinical factors. Flynn scoring will be applied to evaluate improvements in elbow function following battle rope training for children with post-traumatic elbow contracture.

CONTACTS AND LOCATIONS:
Overall Officials: Azlfa Karim, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beck CM, Gluck MJ, Zhang Y, McGough JD, Reizner W, Rubin TA, Hausman MR. Outcomes of Arthroscopic Elbow Contracture Release: Improvement for Severe Prosupination and Flexion Contracture. Arthroscopy. 2022 Feb;38(2):315-322. doi: 10.1016/j.arthro.2021.07.020. Epub 2021 Jul 27. PMID 34329701